CLINICAL TRIAL: NCT03120559
Title: Can we Still Save Dental Floss? Improving Dental Floss Adherence and Gingival Health With SMS and an Innovative Floss Holder in a Randomized Controlled Trial
Brief Title: Improving Dental Floss Adherence and Gingival Health With SMS and an Innovative Floss Holder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Responsible Party: Principal Investigator, Mario Rui Araújo, Master in Health Psychology, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07/2014
Record Dates: First submitted 2017-04-10; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Behavior; Gingivitis
Keywords: Gingivitis; SMS; Dental floss; behavior change; HAPA
MeSH Terms: conditions — Behavior; Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The researcher was blind to the patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The dental consultation was the same for all the groups.
  1. - Examination and diagnosis (15 min).
  2. - Motivation, discussion about desired outcomes and treatment needs followed by instrumentation (scaling, polishing) (30 min).
  3. - Therapeutic goals, therapeutic strategies, teaching skills (brushing and interproximal control with regular waxed floss at the Control group) and scheduling of the follow-up appointment (15 min).
  They were properly organized in accordance with the features of each patient, such as their gingival condition, gingivitis perception, habits and expectancies concerning the treatment. The consultation time was 60 minutes and also included specific behavior change techniques, such as reinforcement, goal-setting, and feedback.
- NFH - New Floss Holder (Other): The dental consultation was the same for all the groups. They were properly organized in accordance with the features of each patient, such as their gingival condition, gingivitis perception, habits and expectancies concerning the treatment. The consultation time was 60 minutes and also included specific behavior change techniques, such as reinforcement, goal-setting, and feedback. New Floss Holder - Gum Chucks
  Interventions: Device: New Floss Holder - Gum Chucks
- New Floss Holder and Short Messages (Other): The dental consultation was the same for all the groups. They were properly organized in accordance with the features of each patient, such as their gingival condition, gingivitis perception, habits and expectancies concerning the treatment. The Intervention time was 60 minutes and also included behavior change techniques, such as reinforcement, goal-setting, and feedback. Participants in the NFH/SMS group further received a total of 16 messages (SMS).
  New Floss Holder - Gum Chucks/SMS
  Interventions: Device: New Floss Holder - Gum Chucks/SMS

INTERVENTIONS:
Device: New Floss Holder - Gum Chucks — Dental inter-proximal control with GumChucks floss holder
  Arms: NFH - New Floss Holder
Device: New Floss Holder - Gum Chucks/SMS — Dental inter-proximal control with GumChucks floss holder and receiving 16 SMS during first 4 months.
  Arms: New Floss Holder and Short Messages

SUMMARY:
This study proposes to evaluate the effects of using a new floss holder (GumChuck) and the use of text messages during supportive periodontal therapy, on the psychological, behavioral and clinical parameters of patients with gingivitis, outlined by evidence and a theory-based framework.

DETAILED DESCRIPTION:
Despite evidence on the benefits of controlling dental biofilm for preventing gingivitis, patients have difficulty complying. Floss holder devices and SMS may be useful in enhancing both the frequency and effectiveness of dental hygiene behaviors, by increasing patients' motivation and self-regulation efforts, but scarce scientific literature supporting their worth in controlling gingivitis and the underlying psychological processes is currently available.

ELIGIBILITY:
Inclusion Criteria:

* Gingivitis BOMP > 0.5
* 20 teeth (minimum 5 per quadrant)
* > 18 years old

Exclusion Criteria:

* periodontitis (pockets >3),
* smoking,
* orthodontics,
* pregnancy
* removable partial dentures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2016-03-30 (Actual)

PRIMARY OUTCOMES:
Change from BOMP (Bleeding on Marginal Probing) at 4 months | Baseline & 4 months
  Gingival bleeding Index

SECONDARY OUTCOMES:
HAPA behavioral variables questionnaire. | Baseline & 4 months
  Assessment of HAPA variables (same 5 points Likert scale for each of the variables)
SMS opinion questionnaire | 4 months
  Opinion about receiving SMS and how can it influence the appointment
Self-report Dental Hygiene Behaviors questionnaire. | Baseline & 4 months
  Level of tooth-brushing and dental floss frequency.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van der Weijden GA, Timmerman MF, Nijboer A, Reijerse E, Van der Velden U. Comparison of different approaches to assess bleeding on probing as indicators of gingivitis. J Clin Periodontol. 1994 Oct;21(9):589-94. doi: 10.1111/j.1600-051x.1994.tb00748.x. PMID 7806674